CLINICAL TRIAL: NCT04456140
Title: Inherit - A Trial of Pro-Active Genetic Testing in Cancer Patients at St. Vincent's Mayo Clinic Embedded Cancer Center
Brief Title: Pro-Active Genetic Testing in Patients With Solid Tumors, Inherit Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Niloy Jewel (Jewel) Samadder, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-011472; NCI-2020-04429 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-011472 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2020-06-24; First posted 2020-07-02 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Breast Carcinoma; Digestive System Neoplasm; Malignant Brain Neoplasm; Malignant Central Nervous System Neoplasm; Malignant Female Reproductive System Neoplasm; Malignant Genitourinary System Neoplasm; Malignant Head and Neck Neoplasm; Malignant Musculoskeletal Neoplasm; Malignant Solid Neoplasm; Metastatic Malignant Neoplasm of Unknown Primary; Skin Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Digestive System Neoplasms; Brain Neoplasms; Central Nervous System Neoplasms; Urogenital Neoplasms; Head and Neck Neoplasms; Neoplasms, Unknown Primary | interventions — Genetic Counseling; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (pre-genetic test counseling, genetic testing) (Experimental): Patients watch a pre-recorded genetic counseling video and those who consent to genetic testing undergo collection of blood samples. Patients also complete surveys over 5-15 minutes each prior to receiving their genetic test results and following the receipt of genetic test results.
  Interventions: Procedure: Biospecimen Collection; Other: Genetic Counseling; Other: Genetic Testing; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
Other: Genetic Counseling — Watch pre-test genetic counseling video
Other: Genetic Testing — Undergo genetic testing
  Other Names: genetic analysis; Genetic Examination; Genetic Test
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase I trial collects blood samples to investigate the prevalence of changes in genes (genetic mutations) in solid tumor patient populations seeking care at Mayo Clinic Embedded Cancer Center at St. Vincent's Riverside. This may help doctors better understand and/or treat others who have genetic mutations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the prevalence of genetic mutations in cancer patients seeking care at the Mayo Clinic Cancer Center at St. Vincent's Riverside in Jacksonville, Florida.

SECONDARY OBJECTIVES:

I. Perform a chart review to assess the impact of genetic testing as part of standard of oncology care:

Ia. Determine differences in germline mutation detection in these patients as compared to traditional guideline (National Comprehensive Cancer Network [NCCN]) based approach for genetic evaluation.

Ib. Determine the percentage of relatives of mutation positive probands undergoing family variant testing within a 3 month window of return of testing results.

Ic. Assess patient experience and barriers to care with a genetic service line via survey measures.

Id. Develop a biorepository of samples (blood) from cancer patients participating in this protocol.

OUTLINE:

Patients watch a pre-recorded genetic counseling video and those who consent to genetic testing undergo collection of blood samples. Patients also complete surveys over 5-15 minutes each prior to receiving their genetic test results and following the receipt of genetic test results.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with any solid tumor cancer (stages 1-4) including, but not limited to, gastrointestinal, breast, gynecological, genitourinary, skin, central nervous system (CNS)/brain, head/neck, musculoskeletal or cancer of unknown primary
* Blood collection is feasible (health, access and/or tolerability) for requested blood sample(s)
* Individuals have agreed to participate and signed the study informed consent form

Exclusion Criteria:

* Individuals who do not meet study inclusion criteria
* Individuals with an active hematologic malignancy
* Patients who have had prior germline genetic testing involving a 40+ gene panel within the last 24 months at Mayo Clinic or St Vincent's Healthcare and available for review by the research coordinator at time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Prevalence of pathogenic germline mutations | Up to 3 months
  Will be assessed by each cancer site, age (< 60 years old versus [vs.] >= 60 years old), and stage (early vs. advanced) via descriptive statistics.
Difference between prevalence of positive pathogenic germline mutations | Up to 3 months
  Will be assessed by cancer sites, age of diagnosis, and stage of diagnosis using logistic regression analysis across all cancer site groups, and pairwise post-hoc analyses using Tukey's correction for multiple comparisons across pairs of cancer sites, and chi-square tests of differences between age and stage groups.
Rate of mutation detection | Up to 3 months
  Will be compared via genetic testing to clinical practice guidelines of traditional family history criteria within cancer site, age, and stage using logistic regression and pairwise post-hoc analyses as needed.
Incidence rate of germline pathogenic genetic mutations in cancer patients seen at St Vincent's and uptake rate of cascade testing in families | Up to 3 months
  Assessed using logistic regression
Incidence rate of germline pathogenic genetic mutations in cancer patients seen at St Vincent's and uptake rate of cascade testing in families | Up to 3 months
  Assessed using pairwise post-hoc analyses

SECONDARY OUTCOMES:
Differences in survey responses between patient groups | Up to 3 months
  Patients will be grouped by genetic test result (positive vs. negative), age (< 60 years old vs. >= 60 years old), stage (early vs. advanced), and over time (enrollment vs. after test results are received).

CONTACTS AND LOCATIONS:
Overall Officials: Niloy J Samadder, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida